CLINICAL TRIAL: NCT05116787
Title: A Randomized, Double-Blind, Multicenter, Placebo-Controlled, Parallel-Group Study to Evaluate the Efficacy, Safety, and Tolerability of Oral BCX9930 Monotherapy for the Treatment of Paroxysmal Nocturnal Hemoglobinuria
Brief Title: BCX9930 for the Treatment of Paroxysmal Nocturnal Hemoglobinuria (PNH) in Participants Not Receiving Other Complement Inhibitor Therapy
Acronym: REDEEM-2
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: BioCryst Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BCX9930-203; 2020-004403-14 (EudraCT Number)
Record Dates: First submitted 2021-11-02; First posted 2021-11-11 (Actual); Results first posted 2025-01-03 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2024-12

CONDITIONS: Paroxysmal Nocturnal Hemoglobinuria (PNH)
Keywords: BCX9930; factor D inhibitor; proximal complement inhibitor; oral therapy; paroxysmal nocturnal hemoglobinuria
MeSH Terms: conditions — Hemoglobinuria, Paroxysmal

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- BCX9930/BCX9930 (Experimental): Participants received BCX9930 monotherapy in double blind manner (Part 1) for 12 weeks, then in an open-label manner for the remainder of the study (Part 2). After the sponsor decided to halt enrolment in the study permanently and terminate the study, participants on blinded study treatment were switched to open-label BCX9930 prior to Week 12. Initially participants were to receive BCX9930 500 mg twice daily (BID) orally. Per protocol amendment, participants who previously received 500 mg BID and remained on study treatment were dose adjusted to 400 mg BID. For all newly enrolled participants, at the initiation of BCX9930 dosing, participants were administered a dose of 200 mg BID for the first 14 days of treatment before increasing to 400 mg BID. The maximum treatment duration in Part 1 was 12 weeks. The overall maximum duration on BCX9930 was 378 days.
  Interventions: Drug: BCX9930 monotherapy
- Placebo/BCX9930 (Placebo Comparator): Participants received BCX9930 matching placebo in double blind manner for 12 weeks (Part 1). After the sponsor decided to halt enrolment in the study permanently and terminate the study, participants switched to open-label BCX9930 monotherapy (Part 2) prior to Week 12, if earlier. The maximum duration on Placebo in Part 1 was 12 weeks. The maximum treatment duration on BCX9930 was 281 days.
  Interventions: Drug: Placebo; Drug: BCX9930 monotherapy

INTERVENTIONS:
Drug: Placebo — Administered orally twice daily
  Arms: Placebo/BCX9930
Drug: BCX9930 monotherapy — Administered orally twice daily

SUMMARY:
The purpose of this study was to determine the efficacy and safety of BCX9930 monotherapy for the treatment of adult participants with PNH not currently receiving complement inhibitor therapy.

DETAILED DESCRIPTION:
This was a randomized, placebo-controlled, double-blind, parallel-group, 2-part study. Parts 1 and 2 was to be conducted in the same participants.

Part 1 of the study was designed to evaluate the efficacy, safety, and tolerability of treatment with oral BCX9930 monotherapy for 12 weeks versus placebo in participants with PNH who were not currently receiving treatment with complement inhibitor therapy. Participants were randomized to receive BCX9930 or placebo under double blind conditions for the 12-week randomized treatment period. The primary efficacy and safety analyses were based on Part 1.

Part 2 of the study was designed to evaluate the long-term safety, tolerability, and effectiveness of open-label BCX9930 monotherapy when administered through Week 52. All participants in Part 2 received BCX9930. Participants who were randomized to BCX9930 monotherapy in Part 1 continued to receive BCX9930 in Part 2. Participants who were randomized to placebo in Part 1 discontinued that therapy at the Week 12 visit and received BCX9930 in Part 2.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged ≥ 18 years old
* Body weight ≥ 40 kg
* Documented diagnosis of PNH
* No complement inhibitor therapy for ≥ 12 months prior to screening
* Contraindication to or no access to approved (C3 or C5) complement inhibitor therapies
* Documentation of current vaccinations against Neisseria meningitidis and Streptococcus pneumoniae or willingness to start vaccination series
* At screening: PNH clone of ≥ 10%, hemoglobin ≤ 10.5 g/dL and lactate dehydrogenase ≥ 2 × upper limit of normal

Exclusion Criteria:

* Known history of or existing diagnosis of hereditary complement deficiency
* History of hematopoietic cell transplant or solid organ transplant or anticipated candidate for transplantation
* Myocardial infarction or cerebrovascular accident within 30 days prior to screening, or current and uncontrolled clinically significant cardiovascular or cerebrovascular condition
* History of malignancy within 5 years prior to the screening visit
* Active bacterial, viral, or fungal infection or any other serious infection within 14 days prior to screening
* Treatment with anti-thymocyte globulin within 180 days prior to screening
* Initiation of treatment with an erythrocyte or platelet growth factor, or danazol within 28 days prior to screening
* Receiving iron supplementation with an unstable dose in the 28 days prior to screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2021-10-26 (Actual); Primary Completion 2023-09-18 (Actual); Study Completion 2023-09-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David J Kuter, MD, DPhil, Principal Investigator — Massachusetts General Hospital
Locations (5):
- Investigative Site, Ampang, Malaysia
- South Africa (3):
  - Investigative Site, Bloemfontein
  - Investigative Site, Cape Town
  - Investigative Site, Pretoria
- InvestigativeSite, Daejeon, South Korea

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted in Malaysia, South Africa, and Korea.
Pre-assignment Details: A total 12 participants were randomized and treated.
Groups:
- BCX9930/BCX9930: Participants received BCX9930 monotherapy in double blind (DB) manner (Part 1) for 12 weeks, then in an open-label manner for the remainder of the study (Part 2). After the sponsor decided to halt enrolment in the study permanently and terminate the study, participants on blinded study treatment were switched to open-label BCX9930 prior to Week 12. Initially participants were to receive BCX9930 500 mg twice daily (BID), orally. Per protocol amendment, participants who previously received 500 mg BID and remained on study treatment were dose adjusted to 400 mg BID. For all newly enrolled participants, at the initiation of BCX9930 dosing, participants were administered a dose of 200 mg BID for the first 14 days of treatment before increasing to 400 mg BID. The maximum treatment duration in Part 1 was 12 weeks. The overall maximum duration on BCX9930 was 378 days.
Period: Part 1:DB Phase (up to 12 Weeks)
Arm/Group | BCX9930/BCX9930 | Placebo/BCX9930
Started | 10 | 2
Completed | 8 | 1
Not Completed | 2 | 1
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Pregnancy | 1 | 0
Not completed — Adverse Event | 1 | 0
Period: Part 2:Open-label Phase (up to 52 Weeks)
Arm/Group | BCX9930/BCX9930 | Placebo/BCX9930
Started | 8 | 1
Completed | 4 | 1
Not Completed | 4 | 0
Not completed — Miscellaneous | 4 | 0

BASELINE CHARACTERISTICS:
Population: The safety population included all participants who received at least 1 dose of study drug, whether placebo or BCX9930. Therefore, BCX9930 group included participants who received BCX9930 throughout the study and placebo group included data for participants who received placebo initially and then switched to BCX9930.
Groups:
- BCX9930/BCX9930: Participants received BCX9930 monotherapy in double blind manner (Part 1) for 12 weeks, then in an open-label manner for the remainder of the study (Part 2). After the sponsor decided to halt enrolment in the study permanently and terminate the study, participants on blinded study treatment were switched to open-label BCX9930 prior to Week 12. Initially participants were to receive BCX9930 500 mg BID orally. Per protocol amendment, participants who previously received 500 mg BID and remained on study treatment were dose adjusted to 400 mg BID. For all newly enrolled participants, at the initiation of BCX9930 dosing, participants were administered a dose of 200 mg BID for the first 14 days of treatment before increasing to 400 mg BID. The maximum treatment duration in Part 1 was 12 weeks. The overall maximum duration on BCX9930 was 378 days.
- Placebo/BCX9930: Participants received BCX9930 matching placebo in double blind manner for 12 weeks (Part 1). After the sponsor decided to halt enrolment in the study permanently and terminate the study, participants switched to open-label BCX9930 monotherapy (Part 2) prior to Week 12, if earlier. The maximum treatment duration in Part 1 was 12 weeks. The maximum duration on Placebo in Part 1 was 12 weeks. The maximum treatment duration on BCX9930 was 281 days.
- Total: Total of all reporting groups
Arm/Group | BCX9930/BCX9930 | Placebo/BCX9930 | Total
Number analyzed (Participants) | 10 | 2 | 12
Age, Continuous [Mean (Standard Deviation); unit: Years] | 37.8 (12.70) | 37.0 (9.90) | 37.7 (11.87)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 2 | 8
  Male | 4 | 0 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 10 | 2 | 12
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 2 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 0 | 7
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Change From Baseline in Hemoglobin at Week 12
Time Frame: Baseline, Week 12
Population: Participants in the All Subjects as Treated (ASaT) population (all participants who received at least 1 dose of study drug and had a post baseline laboratory assessment) in Part 1 were analyzed.
Measure: Mean (Standard Deviation); unit: grams per deciliter (g/dL)
Groups:
- BCX9930: Participants received BCX9930 monotherapy in double blind manner (Part 1) for 12 weeks. Initially participants were to receive BCX9930 500 mg BID orally. Per protocol amendment, participants who previously received 500 mg BID and remained on study treatment were dose adjusted to 400 mg BID. For all newly enrolled participants, at the initiation of BCX9930 dosing, participants were administered a dose of 200 mg BID for the first 14 days of treatment before increasing to 400 mg BID.
- Placebo: Participants received BCX9930 matching placebo in double blind manner for 12 weeks (Part 1).
Arm/Group | BCX9930 | Placebo
Number analyzed (Participants) | 10 | 2
grams per deciliter (g/dL)
  Baseline | 8.49 (1.556) | 9.48 (1.721)
  Change at Week 12 | 2.23 (2.146) | -1.23 (0.330)

2. Secondary Outcome: Part 1: Number of Participants Who Were Transfusion-free
Description: The number of participants who did not receive any transfusions (packed red blood cells [pRBCs] or whole blood) during the period of interest were reported. Participants who were transfusion free were defined for each treatment group as the number of participants who did not receive any transfusions (pRBCs or whole blood) during the period of interest from the start to the end, inclusive, divided by the total number of participants in that treatment group at the start of the period of interest. Participants who (1) discontinued treatment prior to Week 12, or (2) did not receive a transfusion during the period of interest despite recording a Hemoglobin (Hb) value ≤ 9 g/dL with symptoms assessed by the investigator as warranting transfusion or a Hb value ≤ 7 g/dL regardless of symptoms were not considered transfusion free.
Time Frame: From Week 4 to Week 12
Population: Participants in the ASaT population in Part 1 were analyzed.
Measure: Count of Participants; unit: Participants
Groups:
- BCX9930: Participants received BCX9930 monotherapy in double blind manner (Part 1). Initially participants were to receive BCX9930 500 mg BID orally. Per protocol amendment, participants who previously received 500 mg BID and remained on study treatment were dose adjusted to 400 mg BID. For all newly enrolled participants, at the initiation of BCX9930 dosing, participants were administered a dose of 200 mg BID for the first 14 days of treatment before increasing to 400 mg BID.
Arm/Group | BCX9930 | Placebo
Number analyzed (Participants) | 10 | 2
Participants | 8 | 1

3. Secondary Outcome: Part 1: Number of Units of pRBCs Transfused
Time Frame: From Week 4 to Week 12
Population: Participants in the ASaT population in Part 1 were analyzed.
Measure: Number; unit: units of pRBCs
Arm/Group | BCX9930 | Placebo
Number analyzed (Participants) | 10 | 2
units of pRBCs | 1 | 0

4. Secondary Outcome: Part 1: Percent Change From Baseline in Lactate Dehydrogenase
Time Frame: Baseline, Week 12
Population: Participants in the ASaT population in Part 1 were analyzed.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | BCX9930 | Placebo
Number analyzed (Participants) | 10 | 2
percent change | -69.8 (26.00) | 9.1 (45.47)

5. Secondary Outcome: Part 1: Change From Baseline in Functional Assessment of Chronic Illness Therapy (FACIT)-Fatigue Scale Score
Description: The FACIT-Fatigue scale questionnaire was used to determine the level of fatigue experienced by participants. This questionnaire was a 13-item measure that assessed self-reported fatigue and its impact upon daily activities and function. Item scores ranged from 0 ("not at all") to 4 ("very much"), and the total score ranged from 0 to 52, with higher scores indicating greater quality of life.
Time Frame: Baseline, Week 12
Population: Participants in the ASaT population in Part 1 with available data were analyzed.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | BCX9930 | Placebo
Number analyzed (Participants) | 9 | 2
Scores on a scale
  Baseline | 34.3 (13.47) | 13.0 (8.49)
  Change at Week 12: number analyzed (Participants) | 8 | 2
  Change at Week 12 | -2.3 (13.48) | -2.0 (0.00)

6. Secondary Outcome: Part 1: Percentage (%) Reduction in the Rate of pRBC Units Transfused
Description: The rate of pRBC units transfused from Week 4 to Week 12 was calculated and compared to the rate of pRBC units transfused prestudy during the 12 months prior to screening. The percent reduction in rate of pRBC units transfused was the percent difference in rate relative to the prestudy rate, calculated as: (current rate - prestudy rate)/prestudy rate * 100%. Total rate among all participants was evaluated here. Rate of pRBC units transfusion was defined as the percentage of participants who received pRBC transfusions.
Time Frame: Prestudy (12 months prior to screening) and from Week 4 to Week 12
Population: Participants in the ASaT population in Part 1 were analyzed.
Measure: Number; unit: percent reduction
Arm/Group | BCX9930 | Placebo
Number analyzed (Participants) | 10 | 2
percent reduction | 89 | 100

7. Secondary Outcome: Part 1: Number of Participants With Hemoglobin ≥ 12 g/dL
Time Frame: At Week 12
Population: Participants in the ASaT population in Part 1 were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | BCX9930 | Placebo
Number analyzed (Participants) | 10 | 2
Participants | 2 | 0

8. Secondary Outcome: Part 1: Number of Participants Achieving Hemoglobin Stabilization
Description: Hemoglobin stabilization was defined as the participants who avoided 2 g/dL or greater decrease in hemoglobin in the absence of transfusion from Week 4 to Week 12.
Time Frame: From Week 4 to Week 12
Population: Participants in the ASaT population in Part 1 with available data were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | BCX9930 | Placebo
Number analyzed (Participants) | 8 | 2
Participants | 8 | 2

9. Secondary Outcome: Part 1: Change From Baseline in Total Paroxysmal Nocturnal Hemoglobinuria (PNH) Red Blood Cell (RBC) Clone Size
Description: The total PNH RBC clone size refers to the percentage of PNH affected (ie, Type 2 and 3) RBC cells within the total RBC population.
Time Frame: Baseline, Week 12
Population: Participants in the ASaT population Part 1 were analyzed.
Measure: Mean (Standard Deviation); unit: % of PNH-RBC within total RBC population
Arm/Group | BCX9930 | Placebo
Number analyzed (Participants) | 10 | 2
% of PNH-RBC within total RBC population
  Baseline | 50.16 (30.386) | 33.72 (3.765)
  Change at Week 12 | 30.76 (25.925) | -2.15 (0.032)

10. Secondary Outcome: Part 1: Change From Baseline in Ratio of Total PNH RBC Clone Size to PNH White Blood Cell (WBC) Clone Size
Description: The total PNH RBC clone size refers to the percentage of PNH-affected (i.e, Type 2 and 3) RBCs within the total RBC population. The PNH WBC clone size refers to the percentage of PNH-affected WBCs within the total WBC population. The ratio of total PNH RBC clone size to PNH WBC clone size = ratio of percent total PNH RBCs / percent PNH WBCs.
Time Frame: Baseline, Week 12
Population: Participants in the ASaT population in Part 1 with available data were analyzed.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | BCX9930 | Placebo
Number analyzed (Participants) | 7 | 1
ratio
  Baseline | 0.6425 (0.28016) | 0.6860
  Change at Week 12 | 0.2905 (0.26628) | -0.3052

11. Secondary Outcome: Part 1: Change From Baseline in Absolute Reticulocyte Count (ARC)
Time Frame: Baseline, Week 12
Population: Participants in the ASaT population in Part 1 with available data were analyzed.
Measure: Mean (Standard Deviation); unit: 10^9 cells/microliter (μL)
Arm/Group | BCX9930 | Placebo
Number analyzed (Participants) | 10 | 2
10^9 cells/microliter (μL)
  Baseline | 200.01 (81.094) | 261.47 (13.529)
  Change at Week 12: number analyzed (Participants) | 9 | 1
  Change at Week 12 | -111.01 (80.799) | -21.43

12. Secondary Outcome: Part 1: Number of Participants With ARC in the Normal Range
Description: Number of participants with ARC in the normal range (50 - 100 x 10^9 cells/L) were reported.
Time Frame: Week 12
Population: Participants in the ASaT population in Part 1 with available data were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | BCX9930 | Placebo
Number analyzed (Participants) | 9 | 1
Participants | 5 | 0

13. Secondary Outcome: Part 1: Change From Baseline in Haptoglobin
Time Frame: Baseline, Week 12
Population: Participants in the ASaT population in Part 1 were analyzed.
Measure: Mean (Standard Deviation); unit: grams per liter (g/L)
Arm/Group | BCX9930 | Placebo
Number analyzed (Participants) | 10 | 2
grams per liter (g/L)
  Baseline | 0.182 (0.0711) | 0.195 (0.1485)
  Change at Week 12 | 0.493 (0.6948) | 0.000 (0.0000)

14. Secondary Outcome: Part 1: Number of Participants With Haptoglobin ≥ Lower Limit of Normal (LLN) Reference Range
Description: Number of participants with haptoglobin ≥ LLN Reference Range (≥0.3 g/L) were reported.
Time Frame: Week 12
Population: Participants in the ASaT population in Part 1 were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | BCX9930 | Placebo
Number analyzed (Participants) | 10 | 2
Participants | 5 | 1

15. Secondary Outcome: Part 1: Change From Baseline in Total Bilirubin
Time Frame: Baseline, Week 12
Population: Participants in the ASaT population in Part 1 were analyzed.
Measure: Mean (Standard Deviation); unit: milligram per deciliter (mg/dL)
Arm/Group | BCX9930 | Placebo
Number analyzed (Participants) | 10 | 2
milligram per deciliter (mg/dL)
  Change at Week 12 | -0.97 (1.706) | 0.80 (0.283)
  Baseline | 1.66 (1.944) | 3.45 (2.475)

16. Secondary Outcome: Part 1: Change From Baseline in Aspartate Aminotransferase (AST)
Time Frame: Baseline, Week 12
Population: Participants in the ASaT population in Part 1 were analyzed.
Measure: Mean (Standard Deviation); unit: Units per liter (U/L)
Arm/Group | BCX9930 | Placebo
Number analyzed (Participants) | 10 | 2
Units per liter (U/L)
  Baseline | 107.43 (71.295) | 83.60 (6.505)
  Change at Week 12 | -68.83 (58.333) | 13.00 (36.487)

ADVERSE EVENTS:
Time Frame: From Day 1 up to 408 days
Description: The safety population included all participants who received at least 1 dose of study drug, whether placebo or BCX9930.
Groups:
- BCX9930/BCX9930: Participants received BCX9930 monotherapy in double blind manner (Part 1) for 12 weeks, then in an open-label manner for the remainder of the study (Part 2). After the sponsor decided to halt enrolment in the study permanently and terminate the study, participants on blinded study treatment were switched to open-label BCX9930 prior to Week 12. Initially participants were to receive BCX9930 500 mg BID orally. Per protocol amendment, participants who previously received 500 mg BID and remained on study treatment were dose adjusted to 400 mg BID. For all newly enrolled participants, at the initiation of BCX9930 dosing, participants were administered a dose of 200 mg BID for the first 14 days of treatment before increasing to 400 mg BID. The maximum treatment duration was 378 days.
- BCX9930 After Placebo: Participants who were initially randomized to placebo group received BCX9930 monotherapy in open label manner, if they had completed Week 12 on placebo, or earlier after the sponsor decided to halt enrolment in the study permanently and terminate the study. Initially participants were to receive BCX9930 500 mg BID orally. Per protocol amendment, participants who previously received 500 mg BID and remained on study treatment were dose adjusted to 400 mg BID. For all newly enrolled participants, at the initiation of BCX9930 dosing, participants were administered a dose of 200 mg BID for the first 14 days of treatment before increasing to 400 mg BID. The maximum treatment duration was 281 days.
Arm/Group | BCX9930/BCX9930 | Placebo | BCX9930 After Placebo
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/2 | 0/1
Serious Adverse Events (participants affected / at risk) | 5/10 | 1/2 | 1/1
Other Adverse Events (participants affected / at risk) | 10/10 | 2/2 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BCX9930/BCX9930 (N=10) | Placebo (N=2) | BCX9930 After Placebo (N=1)
Enterovirus infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia fungal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Tuberculosis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Breakthrough haemolysis (Blood and lymphatic system disorders) | 1 (2) | 0 (0) | 0 (0)
Budd-Chiari syndrome (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | BCX9930/BCX9930 (N=10) | Placebo (N=2) | BCX9930 After Placebo (N=1)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 0 (0) | 1 (2)
Abdominal pain (Gastrointestinal disorders) | 3 (4) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Varices oesophageal (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Abdominal tenderness (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0)
Gastric varices (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 6 (8) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 (5) | 0 (0) | 0 (0)
Alopecia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Rash papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 4 (5) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pulmonary tuberculosis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Tonsillitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 3 (4) | 1 (1) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 1 (1) | 0 (0) | 0 (0)
Malaise (General disorders) | 1 (1) | 0 (0) | 0 (0)
Peripheral swelling (General disorders) | 0 (0) | 1 (1) | 0 (0)
Swelling face (General disorders) | 1 (1) | 0 (0) | 0 (0)
Vaccination site pruritus (General disorders) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (4) | 0 (0) | 1 (1)
Arthritis reactive (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Joint stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Periarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Breakthrough haemolysis (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0)
Haemolysis (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (2)
Headache (Nervous system disorders) | 4 (6) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Blood uric acid increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Serum ferritin decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Weight increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Haemoglobinuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Nephropathy (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Breast pain (Reproductive system and breast disorders) | 1/6 (1) | 0 (0) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 1/6 (2) | 0 (0) | 0 (0)
Heavy menstrual bleeding (Reproductive system and breast disorders) | 1/6 (2) | 0 (0) | 0 (0)
Menometrorrhagia (Reproductive system and breast disorders) | 0/6 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 1 (2) | 0 (0) | 0 (0)
Jaundice (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
The sponsor decided to terminate the development program (including this study).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2022-08-01): https://cdn.clinicaltrials.gov/large-docs/87/NCT05116787/Prot_000.pdf
  • Statistical Analysis Plan (2023-10-04): https://cdn.clinicaltrials.gov/large-docs/87/NCT05116787/SAP_001.pdf